CLINICAL TRIAL: NCT01702428
Title: Consistency Study of GSK Biologicals' Measles-mumps-rubella (MMR) Vaccine (209762) (Priorix) Comparing Immunogenicity and Safety to Merck & Co., Inc.'s MMR Vaccine (M-M-R II), in Healthy Children 12 to 15 Months of Age
Brief Title: Consistency Study of GlaxoSmithKline (GSK) Biologicals' MMR Vaccine (209762) (Priorix) Comparing Immunogenicity and Safety to Merck & Co., Inc.'s MMR Vaccine (M-M-R II), in Children 12 to 15 Months of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 115648; 2011-004891-12 (EudraCT Number)
Record Dates: First submitted 2012-10-04; First posted 2012-10-08 (Estimated); Results first posted 2018-06-28 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Rubella; Measles; Mumps
Keywords: Safety; Consistency study; Measles, mumps and rubella diseases; Healthy children; Immunogenicity
MeSH Terms: conditions — Rubella; Measles; Mumps | interventions — Measles-Mumps-Rubella Vaccine; Rubella Vaccine; Chickenpox Vaccine; Hepatitis A Vaccines; 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- INV_MMR_L1 Group (Experimental): Subjects receive 1 dose of GSK's candidate combined measles, mumps and rubella (MMR) investigational vaccine (INV_MMR) Lot 1 (L1) co-administered with VV and HAV vaccines at Visit 1 (Day 0). All US subjects are also given PCV-13 vaccine. The MMR vaccine is administered subcutaneously in the triceps region of the left arm while the VV vaccine is administered subcutaneously in the triceps region of the right arm. HAV and PCV-13 vaccines are administered intramuscularly in the anterolateral region of the right and left thigh, respectively.
  Interventions: Biological: Priorix; Biological: Varivax; Biological: Havrix; Biological: Prevnar 13
- INV_MMR_L2 Group (Experimental): Subjects receive 1 dose of GSK's candidate combined measles, mumps and rubella (MMR) investigational vaccine (INV_MMR) Lot 2 (L2) co-administered with VV and HAV vaccines at Visit 1 (Day 0). All US subjects are also given PCV-13 vaccine. The MMR vaccine is administered subcutaneously in the triceps region of the left arm while the VV vaccine is administered subcutaneously in the triceps region of the right arm. HAV and PCV-13 vaccines are administered intramuscularly in the anterolateral region of the right and left thigh, respectively.
  Interventions: Biological: Priorix; Biological: Varivax; Biological: Havrix; Biological: Prevnar 13
- INV_MMR_L3 Group (Experimental): Subjects receive 1 dose of GSK's candidate combined measles, mumps and rubella (MMR) investigational vaccine (INV_MMR) Lot 3 (L3) co-administered with VV and HAV vaccines at Visit 1 (Day 0). All US subjects are also given PCV-13 vaccine. The MMR vaccine is administered subcutaneously in the triceps region of the left arm while the VV vaccine is administered subcutaneously in the triceps region of the right arm. HAV and PCV-13 vaccines are administered intramuscularly in the anterolateral region of the right and left thigh, respectively.
  Interventions: Biological: Priorix; Biological: Varivax; Biological: Havrix; Biological: Prevnar 13
- COM_MMR Group (Active Comparator): Subjects receive 1 dose of COM_MMR Lot 1 and Lot 2 co-administered with VV and HAV vaccines at Visit 1 (Day 0). All US subjects are also given PCV-13 vaccine. The MMR vaccine is administered subcutaneously in the triceps region of the left arm while the VV vaccine is administered subcutaneously in the triceps region of the right arm. HAV and PCV-13 vaccines are administered intramuscularly in the anterolateral region of the right and left thigh, respectively. Pooled analysis is conducted for this group.
  Interventions: Biological: M-M-R II; Biological: Varivax; Biological: Havrix; Biological: Prevnar 13

INTERVENTIONS:
Biological: Priorix — Subjects receive 1 dose of MMR vaccine which is administered subcutaneously in the triceps region of the left arm.
  Other Names: GSK Biologicals' live attenuated measles; mumps and rubella vaccine (GSK209762)
  Arms: INV_MMR_L1 Group; INV_MMR_L2 Group; INV_MMR_L3 Group
Biological: M-M-R II — Subjects receive 1 dose of MMR vaccine which is administered subcutaneously in the triceps region of the left arm.
  Arms: COM_MMR Group
Biological: Varivax — Subjects receive 1 dose of VV vaccine which is administered subcutaneously in the triceps region of the right arm.
Biological: Havrix — Subjects receive 1 dose of HAV vaccine which is administered intramuscularly in the anterolateral region of the right thigh.
Biological: Prevnar 13 — US subjects receive 1 dose of PCV-13 vaccine which is administered intramuscularly in the anterolateral region of the left thigh.

SUMMARY:
The purpose of this study is to evaluate consistency in terms of the immune response to three different lots of GSK Biologicals' trivalent MMR vaccine manufactured to target potencies, and compare its immunogenicity to Merck & Co., Inc.'s MMR vaccine, which is approved for use in the United States (US).

DETAILED DESCRIPTION:
This study will evaluate the consistency of the immune response to three different lots of GSK Biologicals' trivalent investigational MMR vaccine (referred to as INV_MMR vaccine, throughout this document) and compare its immunogenicity to the US standard of care comparator vaccine (M-M-R II, Merck and Co., Inc., referred to as COM_MMR throughout this document) in children during their second year of life. The INV_MMR vaccine will be given as one of three consistency lots manufactured to target potencies designated as INV_MMR_L1, INV_MMR_L2 and INV_MMR_L3. The COM_MMR vaccine will be given as one of two lots designated COM_MMR_L1 and COM_MMR_L2 and will be analysed as pooled lots within the study. The MMR vaccine will be co-administered with Varivax (VV), Havrix (HAV) and (in the US sub-cohort only) Prevnar 13 (PCV-13) which are routinely administered to children of this age in the US.

ELIGIBILITY:
Inclusion Criteria:

* Male or female child between 12 and 15 months of age at the time of vaccination.
* The investigator believes that the parent(s) or Legally Acceptable Representative(s) (LAR(s)) of the child, can, and will comply with the requirements of the protocol.
* Written informed consent obtained from the parent(s)/LAR(s) of the child.
* Child is in stable health as determined by investigator's clinical examination and assessment of child's medical history.

For US children only:

• Child that previously received a 3-dose series of Prevnar 13 only (i.e., no doses given as Prevnar/Prevenar), with the last dose at least 60 days prior to study entry.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine(s) during the period starting 30 days before the day of study vaccination (i.e., 30 days prior to Day 0) or planned use during the entire study period.
* Concurrently participating in another clinical study, in which the child has been or will be exposed to an investigational or a non-investigational product.
* Chronic administration of immunosuppressants, or other immune-modifying drugs during the period starting 180 days prior to the first vaccine dose or any planned administration of immunosuppressive and immune-modifying drugs during the entire study.

  * For corticosteroids, this will mean prednisone, ≥0.5 mg/kg/day or equivalent.
  * Inhaled and topical steroids are allowed.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting 30 days prior to study vaccination at Visit 1 and ending at Visit 2. Please Note:

  * Inactivated influenza (Flu) vaccine and Haemophilus influenzae type b conjugate vaccine (Hib) vaccines may be given at any time, including the day of study vaccination (Flu and Hib vaccines must be administered at a different location than the study vaccine/s).
  * Any other age appropriate vaccine may be given starting at Visit 2 and anytime thereafter.
* Administration of immunoglobulins and/or any blood products during the period starting 180 days prior to study vaccination at Visit 1 or planned administration from the date of vaccination through the immunogenicity evaluation at Visit 2.
* History of measles, mumps, rubella, varicella/zoster and/or hepatitis A disease.
* Known exposure to measles, mumps, rubella and/or varicella/zoster during the period starting within 30 days prior to first study vaccination.
* Previous vaccination against measles, mumps, rubella, hepatitis A and/or varicella virus.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines, including hypersensitivity to neomycin, latex or gelatin.
* Blood dyscrasias, leukemia, lymphomas of any type, or other malignant neoplasms affecting the bone marrow or lymphatic systems.
* Acute disease at the time of enrollment. All vaccines can be administered to persons with a minor illness such as diarrhea, mild upper respiratory infection without fever.
* Active untreated tuberculosis based on medical history.
* Any other condition which, in the opinion of the investigator, prevents the child from participating in the study.

For US children only:

* Child that previously received a vaccination with heptavalent Prevnar/Prevenar (prior vaccination should be with 3 doses of Prevnar 13 only).
* Child that previously received a fourth dose of any pneumococcal conjugate vaccine.

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5016 (Actual)
Dates: Start 2012-11-09 (Actual); Primary Completion 2014-11-25 (Actual); Study Completion 2015-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (77):
- United States (59):
  - GSK Investigational Site, Dothan, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Fayetteville, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Daly City, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Hayward, California
  - GSK Investigational Site, Los Gatos, California
  - GSK Investigational Site, Mission Hills, California
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, Pleasanton, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Santa Clara, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Evergreen Park, Illinois
  - GSK Investigational Site, Ames, Iowa
  - GSK Investigational Site, Augusta, Kansas
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Bossier City, Louisiana
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Fall River, Massachusetts
  - GSK Investigational Site, Niles, Michigan
  - GSK Investigational Site, Stevensville, Michigan
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Ithaca, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Hermitage, Pennsylvania
  - GSK Investigational Site, Sellersville, Pennsylvania
  - GSK Investigational Site, Warwick, Rhode Island
  - GSK Investigational Site, Barnwell, South Carolina
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, League City, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Tomball, Texas
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Payson, Utah
  - GSK Investigational Site, Provo, Utah
  - GSK Investigational Site, Roy, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, St. George, Utah
  - GSK Investigational Site, Syracuse, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Falls Church, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Marshfield, Wisconsin
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Finland (9):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- Mexico (2):
  - GSK Investigational Site, Durango
  - GSK Investigational Site, México
- GSK Investigational Site, San Juan, Puerto Rico
- Spain (4):
  - GSK Investigational Site, Castellon
  - GSK Investigational Site, L'Eliana, Valencia
  - GSK Investigational Site, Quart de Poblet, Valencia
  - GSK Investigational Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=19887

REFERENCES:
- [Background] Klein NP, Abu-Elyazeed R, Povey M, Macias Parra M, Diez-Domingo J, Ahonen A, Korhonen T, Tinoco JC, Weiner L, Marshall GS, Silas PE, Sarpong KO, Ramsey KP, Fling JA, Speicher D, Campos M, Munjal I, Peltier C, Vesikari T, Baccarini C, Caplanusi A, Gillard P, Carryn S, Henry O. Immunogenicity and Safety of a Measles-Mumps-Rubella Vaccine Administered as a First Dose to Children Aged 12 to 15 Months: A Phase III, Randomized, Noninferiority, Lot-to-Lot Consistency Study. J Pediatric Infect Dis Soc. 2020 Apr 30;9(2):194-201. doi: 10.1093/jpids/piz010. PMID 30849175

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 13 subjects from 5016 were allocated subject number but no study vaccine was administered. Therefore, the number of subjects started is 5003.
Pre-assignment Details: Sub-cohorts for this study were as follows: • US sub-cohort: Subjects recruited in US and received INV_MMR or COM_MMR co-administered with Varivax (VV), Havrix (HAV) and Prevnar (PCV-13) vaccines at Visit 1 (Day 0). • Non-US sub-cohort: Subjects recruited outside US and received INV_MMR or COM_MMR co-administered with VV and HAV vaccines at Day 0.
Groups:
- INV_MMR_L1 Group: Subjects received 1 dose of GSK's candidate combined measles, mumps and rubella (MMR) investigational vaccine (INV_MMR) Lot 1 (L1) co-administered with VV and HAV vaccines at Visit 1 (Day 0). All US subjects were also given PCV-13 vaccine. The MMR vaccine was administered subcutaneously in the triceps region of the left arm while the VV vaccine was administered subcutaneously in the triceps region of the right arm. HAV and PCV-13 vaccines were administered intramuscularly in the anterolateral region of the right and left thigh, respectively.
- INV_MMR_L2 Group: Subjects received 1 dose of GSK's candidate combined measles, mumps and rubella (MMR) investigational vaccine (INV_MMR) Lot 2 (L2) co-administered with VV and HAV vaccines at Visit 1 (Day 0). All US subjects were also given PCV-13 vaccine. The MMR vaccine was administered subcutaneously in the triceps region of the left arm while the VV vaccine was administered subcutaneously in the triceps region of the right arm. HAV and PCV-13 vaccines were administered intramuscularly in the anterolateral region of the right and left thigh, respectively.
- INV_MMR_L3 Group: Subjects received 1 dose of GSK's candidate combined measles, mumps and rubella (MMR) investigational vaccine (INV_MMR) Lot 3 (L3) co-administered with VV and HAV vaccines at Visit 1 (Day 0). All US subjects were also given PCV-13 vaccine. The MMR vaccine was administered subcutaneously in the triceps region of the left arm while the VV vaccine was administered subcutaneously in the triceps region of the right arm. HAV and PCV-13 vaccines were administered intramuscularly in the anterolateral region of the right and left thigh, respectively.
- COM_MMR Group: Subjects received 1 dose of COM_MMR Lot 1 and Lot 2 co-administered with VV and HAV vaccines at Visit 1 (Day 0). All US subjects were also given PCV-13 vaccine. The MMR vaccine was administered subcutaneously in the triceps region of the left arm while the VV vaccine was administered subcutaneously in the triceps region of the right arm. HAV and PCV-13 vaccines were administered intramuscularly in the anterolateral region of the right and left thigh, respectively. Pooled analysis was conducted for this group.
Period: Overall Study
Arm/Group | INV_MMR_L1 Group | INV_MMR_L2 Group | INV_MMR_L3 Group | COM_MMR Group
Started | 1239 | 1232 | 1243 | 1289
Completed | 1175 | 1162 | 1190 | 1232
Not Completed | 64 | 70 | 53 | 57
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 33 | 41 | 37 | 44
Not completed — Parents cannot assist to site | 1 | 0 | 1 | 0
Not completed — Lost Coverage | 0 | 0 | 0 | 1
Not completed — Lost Health Plan | 3 | 5 | 0 | 2
Not completed — Mother transferred care | 0 | 1 | 0 | 0
Not completed — Parents too busy | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 21 | 23 | 14 | 10

BASELINE CHARACTERISTICS:
Groups:
- INV_MMR_L1 Group: Subjects received 1 dose of INV_MMR_L1 vaccine co-administered with VV and HAV vaccines at Visit 1 (Day 0). All US subjects were also given PCV-13 vaccine. The MMR vaccine was administered subcutaneously in the triceps region of the left arm while the VV vaccine was administered subcutaneously in the triceps region of the right arm. HAV and PCV-13 vaccines were administered intramuscularly in the anterolateral region of the right and left thigh, respectively.
- INV_MMR_L2 Group: Subjects received 1 dose of INV_MMR_L2 vaccine co-administered with VV and HAV vaccines at Visit 1 (Day 0). All US subjects were also given PCV-13 vaccine. The MMR vaccine was administered subcutaneously in the triceps region of the left arm while the VV vaccine was administered subcutaneously in the triceps region of the right arm. HAV and PCV-13 vaccines were administered intramuscularly in the anterolateral region of the right and left thigh, respectively.
- INV_MMR_L3 Group: Subjects received 1 dose of INV_MMR_L3 vaccine co-administered with VV and HAV vaccines at Visit 1 (Day 0). All US subjects were also given PCV-13 vaccine. The MMR vaccine was administered subcutaneously in the triceps region of the left arm while the VV vaccine was administered subcutaneously in the triceps region of the right arm. HAV and PCV-13 vaccines were administered intramuscularly in the anterolateral region of the right and left thigh, respectively.
- Total: Total of all reporting groups
Arm/Group | INV_MMR_L1 Group | INV_MMR_L2 Group | INV_MMR_L3 Group | COM_MMR Group | Total
Number analyzed (Participants) | 1239 | 1232 | 1243 | 1289 | 5003
Age, Continuous [Mean (Standard Deviation); unit: Months] | 12.3 (0.7) | 12.3 (0.7) | 12.3 (0.7) | 12.3 (0.7) | 12.3 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 607 | 594 | 615 | 618 | 2434
  Male | 632 | 638 | 628 | 671 | 2569
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Arabic / North African Heritage | 5 | 6 | 2 | 7 | 20
  Asian - Central/South Asian Heritage | 14 | 6 | 7 | 9 | 36
  Other | 170 | 155 | 162 | 163 | 650
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 5 | 2 | 11
  American Indian or Alaskan Native | 25 | 37 | 33 | 31 | 126
  White - Caucasian / European Heritage | 932 | 938 | 944 | 970 | 3784
  Asian - South East Asian Heritage | 21 | 25 | 21 | 26 | 93
  African Heritage / African American | 60 | 52 | 57 | 70 | 239
  Asian - Japanese Heritage | 1 | 2 | 2 | 1 | 6
  Asian - East Asian Heritage | 8 | 10 | 10 | 10 | 38

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Anti-measles Virus Antibody Concentration Equal to or Above the Cut-off-value
Description: Seroresponse was defined as post-vaccination anti-measles virus antibody concentration ≥200 milli International Unit/Milliliter (mIU/mL) among subjects who were seronegative (antibody concentration <150 mIU/mL) before vaccination. This outcome measure is applicable to reporting groups INV_MMR_L1, INV_MMR_L2 and INV_MMR_L3 as analysis was performed on subjects who received one of the lots of INV_MMR vaccine.
Time Frame: At Day 42
Population: According to protocol (ATP) cohort for immunogenicity included subjects who received at least 1 MMR vaccine, were below the assay cut-off at pre-vaccination & with pre & post dose serology results available for at least 1 antigen of MMR, did not meet any elimination criteria up to Visit 2 blood sample & complied with post dose blood sample schedule
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- INV_MMR _L1 Group: Subjects received 1 dose of INV_MMR_L1 vaccine co-administered with VV and HAV vaccines at Visit 1 (Day 0). All US subjects were also given PCV-13 vaccine. The MMR vaccine was administered subcutaneously in the triceps region of the left arm while the VV vaccine was administered subcutaneously in the triceps region of the right arm. HAV and PCV-13 vaccines were administered intramuscularly in the anterolateral region of the right and left thigh, respectively.
- INV_MMR _L2 Group: Subjects received 1 dose of INV_MMR_L2 vaccine co-administered with VV and HAV vaccines at Visit 1 (Day 0). All US subjects were also given PCV-13 vaccine. The MMR vaccine was administered subcutaneously in the triceps region of the left arm while the VV vaccine was administered subcutaneously in the triceps region of the right arm. HAV and PCV-13 vaccines were administered intramuscularly in the anterolateral region of the right and left thigh, respectively.
- INV_MMR _L3 Group: Subjects received 1 dose of INV_MMR_L3 vaccine co-administered with VV and HAV vaccines at Visit 1 (Day 0). All US subjects were also given PCV-13 vaccine. The MMR vaccine was administered subcutaneously in the triceps region of the left arm while the VV vaccine was administered subcutaneously in the triceps region of the right arm. HAV and PCV-13 vaccines were administered intramuscularly in the anterolateral region of the right and left thigh, respectively.
Arm/Group | INV_MMR _L1 Group | INV_MMR _L2 Group | INV_MMR _L3 Group
Number analyzed (Participants) | 1083 | 1069 | 1096
Percentage of subjects
  Anti-measles ≥ 150 mIU/mL | 98.2 [97.3 to 98.9] | 98.9 [98.0 to 99.4] | 98.1 [97.1 to 98.8]
  Anti-measles ≥ 200 mIU/mL | 98.1 [97.1 to 98.8] | 98.6 [97.7 to 99.2] | 97.8 [96.8 to 98.6]
Statistical Analysis 1: Comparison: INV_MMR _L1 Group vs INV_MMR _L2 Group; Difference between groups (INV_MMR_L1 Group minus INV_MMR_L2 Group) in percentage of subjects with anti-measles antibody concentration ≥200 mIU/mL; Test type: Non-Inferiority or Equivalence — For each pair-wise comparison, the 2-sided 95% confidence interval (CI) on the lot difference in seroresponse rates should be within the [-5%;5%] margin for antibodies to measles virus; Difference in seroresponse rate = -0.54, 95% CI 2-sided [-1.69 to 0.58] — Asymptotic standardized 95% CI for the pair-wise differences in seroresponse
Statistical Analysis 2: Comparison: INV_MMR _L2 Group vs INV_MMR _L3 Group; Difference between groups (INV_MMR_L2 Group minus INV_MMR_L3 Group) in percentage of subjects with anti-measles antibody concentration ≥200 mIU/mL; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in seroresponse rate = 0.79, 95% CI 2-sided [-0.35 to 1.98] — Asymptotic standardized 95% CI for the pair-wise differences in seroresponse
Statistical Analysis 3: Comparison: INV_MMR _L1 Group vs INV_MMR _L3 Group; Difference between groups (INV_MMR_L1 Group minus INV_MMR_L3 Group) in percentage of subjects with anti-measles antibody concentration ≥200 mIU/mL; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in seroresponse rate = 0.25, 95% CI 2-sided [-0.98 to 1.50] — Asymptotic standardized 95% CI for the pair-wise differences in seroresponse

2. Primary Outcome: Anti-measles Virus Antibody Concentrations
Description: Antibody concentrations were expressed as Geometric Mean Concentrations (GMCs) in mIU/mL. This outcome measure is applicable to reporting groups INV_MMR_L1, INV_MMR_L2 and INV_MMR_L3 as analysis was performed on subjects who received one of the lots of INV_MMR vaccine.
Time Frame: At Day 42
Population: ATP cohort for immunogenicity included subjects who received at least 1 MMR vaccine, were below the assay cut-off at pre-vaccination & with pre & post dose serology results available for at least 1 antigen of MMR, did not meet any elimination criteria up to Visit 2 blood sample & complied with post dose blood sample schedule
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | INV_MMR _L1 Group | INV_MMR _L2 Group | INV_MMR _L3 Group
Number analyzed (Participants) | 1083 | 1069 | 1096
mIU/mL | 2970.3 [2813.2 to 3136.2] | 3023.6 [2864.5 to 3191.6] | 3058.3 [2893.9 to 3232.0]
Statistical Analysis 1: Comparison: INV_MMR _L1 Group vs INV_MMR _L2 Group; Adjusted GMC ratio (INV_MMR_L1 Group divided by INV_MMR_L2 Group) for antibodies to measles virus at Day 42; Test type: Non-Inferiority or Equivalence — For each pair-wise comparison, the 2-sided 95% CI on the lot ratio should be within the [0.67;1.5] margin for antibodies to measles; ANOVA; 95% CI for GMC of each INV_MMR lots pair was computed using ANOVA (3 INV_MMR lot groups & country as fixed effects) on log-transformed concentrations; Adjusted GMC ratio = 0.99, 95% CI 2-sided [0.91 to 1.06]
Statistical Analysis 2: Comparison: INV_MMR _L1 Group vs INV_MMR _L3 Group; Adjusted GMC ratio (INV_MMR_L1 Group divided by INV_MMR_L3 Group) for antibodies to measles virus at Day 42; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANOVA; [statistical method as in outcome 2, analysis 1]; Adjusted GMC ratio = 0.97, 95% CI 2-sided [0.90 to 1.05]
Statistical Analysis 3: Comparison: INV_MMR _L1 Group vs INV_MMR _L2 Group; Adjusted GMC ratio (INV_MMR_L2 Group divided by INV_MMR_L1 Group) for antibodies to measles virus at Day 42; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANOVA; [statistical method as in outcome 2, analysis 1]; Adjusted GMC ratio = 1.01, 95% CI 2-sided [0.94 to 1.09]
Statistical Analysis 4: Comparison: INV_MMR _L2 Group vs INV_MMR _L3 Group; Adjusted GMC ratio (INV_MMR_L2 Group divided by INV_MMR_L3 Group) for antibodies to measles virus at Day 42; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANOVA; [statistical method as in outcome 2, analysis 1]; Adjusted GMC ratio = 0.99, 95% CI 2-sided [0.91 to 1.06]
Statistical Analysis 5: Comparison: INV_MMR _L1 Group vs INV_MMR _L3 Group; Adjusted GMC ratio (INV_MMR_L3 Group divided by INV_MMR_L1 Group) for antibodies to measles virus at Day 42; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANOVA; [statistical method as in outcome 2, analysis 1]; Adjusted GMC ratio = 1.03, 95% CI 2-sided [0.95 to 1.11]
Statistical Analysis 6: Comparison: INV_MMR _L2 Group vs INV_MMR _L3 Group; Adjusted GMC ratio (INV_MMR_L3 Group divided by INV_MMR_L2 Group) for antibodies to measles virus at Day 42; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANOVA; [statistical method as in outcome 2, analysis 1]; Adjusted GMC ratio = 1.01, 95% CI 2-sided [0.94 to 1.09]

3. Primary Outcome: Percentage of Subjects With Anti-mumps Virus Antibody Concentration Equal to or Above the Cut-off-value
Description: Seroresponse was defined as post-vaccination anti-mumps virus antibody concentration ≥10 ELISA Unit/Milliliter (EU/mL) among subjects who were seronegative (antibody concentrations <5 EU/mL) before vaccination. This outcome measure is applicable to reporting groups INV_MMR_L1, INV_MMR_L2 and INV_MMR_L3 as analysis was performed on subjects who received one of the lots of INV_MMR vaccine.
Time Frame: At Day 42
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | INV_MMR_L1 Group | INV_MMR_L2 Group | INV_MMR_L3 Group
Number analyzed (Participants) | 1062 | 1047 | 1078
Percentage of subjects
  Anti-mumps ≥ 5 EU/mL | 99.7 [99.2 to 99.9] | 99.3 [98.6 to 99.7] | 99.2 [98.4 to 99.6]
  Anti-mumps ≥ 10 EU/mL | 98.6 [97.7 to 99.2] | 98.6 [97.6 to 99.2] | 98.0 [96.9 to 98.7]
Statistical Analysis 1: Comparison: INV_MMR_L1 Group vs INV_MMR_L2 Group; Difference between groups (INV_MMR_L1 Group minus INV_MMR_L2 Group) in percentage of subjects with anti-mumps antibody concentration ≥10 EU/mL; Test type: Non-Inferiority or Equivalence — For each pair-wise comparison, the 2-sided 95% CI on the lot difference in seroresponse rates should be within the [-5%;5%] margin for antibodies to mumps virus; Difference in seroresponse rate = 0.02, 95% CI 2-sided [-1.05 to 1.09] — Asymptotic standardized 95% CI for the pair-wise differences in seroresponse
Statistical Analysis 2: Comparison: INV_MMR_L1 Group vs INV_MMR_L3 Group; Difference between groups (INV_MMR_L1 Group minus INV_MMR_L3 Group) in percentage of subjects with anti-mumps antibody concentration ≥10 EU/mL; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference in seroresponse rate = 0.63, 95% CI 2-sided [-0.50 to 1.81] — Asymptotic standardized 95% CI for the pair-wise differences in seroresponse
Statistical Analysis 3: Comparison: INV_MMR_L2 Group vs INV_MMR_L3 Group; Difference between groups (INV_MMR_L2 Group minus INV_MMR_L3 Group) in percentage of subjects with anti-mumps antibody concentration ≥10 EU/mL; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference in seroresponse rate = 0.61, 95% CI 2-sided [-0.53 to 1.79] — Asymptotic standardized 95% CI for the pair-wise differences in seroresponse

4. Primary Outcome: Anti-mumps Virus Antibody Concentration
Description: Antibody concentrations were expressed as GMCs in EU/mL. This outcome measure is applicable to reporting groups INV_MMR_L1, INV_MMR_L2 and INV_MMR_L3 as analysis was performed on subjects who received one of the lots of INV_MMR vaccine.
Time Frame: At Day 42
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | INV_MMR_L1 Group | INV_MMR_L2 Group | INV_MMR_L3 Group
Number analyzed (Participants) | 1062 | 1047 | 1078
EU/mL | 71.7 [68.3 to 75.2] | 76.9 [73.2 to 80.8] | 69.0 [65.5 to 72.7]
Statistical Analysis 1: Comparison: INV_MMR_L1 Group vs INV_MMR_L2 Group; Adjusted GMC ratio (INV_MMR_L1 Group divided by INV_MMR_L2 Group) for antibodies to mumps virus at Day 42; Test type: Non-Inferiority or Equivalence — For each pair-wise comparison, the 2-sided 95% CI on the lot ratio should be within the [0.67;1.5] margin for antibodies to mumps; ANOVA; [statistical method as in outcome 2, analysis 1]; Adjusted GMC ratio = 0.93, 95% CI 2-sided [0.87 to 1.00]
Statistical Analysis 2: Comparison: INV_MMR_L1 Group vs INV_MMR_L3 Group; Adjusted GMC ratio (INV_MMR_L1 Group divided by INV_MMR_L3 Group) for antibodies to mumps virus at Day 42; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; ANOVA; [statistical method as in outcome 2, analysis 1]; Adjusted GMC ratio = 1.04, 95% CI 2-sided [0.97 to 1.11]
Statistical Analysis 3: Comparison: INV_MMR_L1 Group vs INV_MMR_L2 Group; Adjusted GMC ratio (INV_MMR_L2 Group divided by INV_MMR_L1 Group) for antibodies to mumps virus at Day 42; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; ANOVA; [statistical method as in outcome 2, analysis 1]; Adjusted GMC ratio = 1.07, 95% CI 2-sided [1.00 to 1.15]
Statistical Analysis 4: Comparison: INV_MMR_L2 Group vs INV_MMR_L3 Group; Adjusted GMC ratio (INV_MMR_L2 Group divided by INV_MMR_L3 Group) for antibodies to mumps virus at Day 42; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; ANOVA; [statistical method as in outcome 2, analysis 1]; Adjusted GMC ratio = 1.11, 95% CI 2-sided [1.04 to 1.19]
Statistical Analysis 5: Comparison: INV_MMR_L1 Group vs INV_MMR_L3 Group; Adjusted GMC ratio (INV_MMR_L3 Group divided by INV_MMR_L1 Group) for antibodies to mumps virus at Day 42; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; ANOVA; [statistical method as in outcome 2, analysis 1]; Adjusted GMC ratio = 0.96, 95% CI 2-sided [0.90 to 1.03]
Statistical Analysis 6: Comparison: INV_MMR_L2 Group vs INV_MMR_L3 Group; Adjusted GMC ratio (INV_MMR_L3 Group divided by INV_MMR_L2 Group) for antibodies to mumps virus at Day 42; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; ANOVA; [statistical method as in outcome 2, analysis 1]; Adjusted GMC ratio = 0.90, 95% CI 2-sided [0.84 to 0.96]

5. Primary Outcome: Percentage of Subjects With Anti-rubella Virus Antibody Concentration Equal to or Above the Cut-off-value
Description: Seroresponse was defined as post-vaccination anti-rubella virus antibody concentration ≥10 International Unit/Milliliter (IU/mL) among subjects who were seronegative (antibody concentrations <4 IU/mL) before vaccination. This outcome measure is applicable to reporting groups INV_MMR_L1, INV_MMR_L2 and INV_MMR_L3 as analysis was performed on subjects who received one of the lots of INV_MMR vaccine.
Time Frame: At Day 42
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | INV_MMR_L1 Group | INV_MMR_L2 Group | INV_MMR_L3 Group
Number analyzed (Participants) | 1083 | 1067 | 1095
Percentage of subjects
  Anti-rubella ≥ 4 IU/mL | 99.4 [98.8 to 99.8] | 99.7 [99.2 to 99.9] | 99.4 [98.7 to 99.7]
  Anti-rubella ≥ 10 IU/mL | 97.2 [96.1 to 98.1] | 97.1 [95.9 to 98.0] | 97.7 [96.6 to 98.5]
Statistical Analysis 1: Comparison: INV_MMR_L1 Group vs INV_MMR_L2 Group; Difference between groups (INV_MMR_L1 Group minus INV_MMR_L2 Group) in percentage of subjects with anti-rubella antibody concentration ≥10 IU/mL; Test type: Non-Inferiority or Equivalence — For each pair-wise comparison, the 2-sided 95% CI on the lot difference in seroresponse rates should be within the [-5%;5%] margin for antibodies to rubella virus; Difference in seroresponse rate = 0.14, 95% CI 2-sided [-1.3 to 1.58] — Asymptotic standardized 95% CI for the pair-wise differences in seroresponse
Statistical Analysis 2: Comparison: INV_MMR_L1 Group vs INV_MMR_L3 Group; Difference between groups (INV_MMR_L1 Group minus INV_MMR_L3 Group) in percentage of subjects with anti-rubella antibody concentration ≥10 IU/mL; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference in seroresponse rate = -0.49, 95% CI 2-sided [-1.86 to 0.86] — Asymptotic standardized 95% CI for the pair-wise differences in seroresponse
Statistical Analysis 3: Comparison: INV_MMR_L2 Group vs INV_MMR_L3 Group; Difference between groups (INV_MMR_L2 Group minus INV_MMR_L3 Group) in percentage of subjects with anti-rubella antibody concentration ≥10 IU/mL; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference in seroresponse rate = -0.62, 95% CI 2-sided [-2.02 to 0.74] — Asymptotic standardized 95% CI for the pair-wise differences in seroresponse

6. Primary Outcome: Anti-rubella Virus Antibody Concentration
Description: Antibody concentrations were expressed as GMCs in IU/mL. This outcome measure is applicable to reporting groups INV_MMR_L1, INV_MMR_L2 and INV_MMR_L3 as analysis was performed on subjects who received one of the lots of INV_MMR vaccine.
Time Frame: At Day 42
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | INV_MMR_L1 Group | INV_MMR_L2 Group | INV_MMR_L3 Group
Number analyzed (Participants) | 1083 | 1067 | 1095
IU/mL | 57.2 [54.4 to 60.1] | 53.1 [50.5 to 55.7] | 57.0 [54.3 to 59.8]
Statistical Analysis 1: Comparison: INV_MMR_L1 Group vs INV_MMR_L2 Group; Adjusted GMC ratio (INV_MMR_L1 Group divided by INV_MMR_L2 Group) for antibodies to rubella virus at Day 42; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANOVA; [statistical method as in outcome 2, analysis 1]; Adjusted GMC ratio = 1.08, 95% CI 2-sided [1.01 to 1.15]
Statistical Analysis 2: Comparison: INV_MMR_L1 Group vs INV_MMR_L3 Group; Adjusted GMC ratio (INV_MMR_L1 Group divided by INV_MMR_L3 Group) for antibodies to rubella virus at Day 42; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANOVA; [statistical method as in outcome 2, analysis 1]; Adjusted GMC ratio = 1.00, 95% CI 2-sided [0.94 to 1.07]
Statistical Analysis 3: Comparison: INV_MMR_L1 Group vs INV_MMR_L2 Group; Adjusted GMC ratio (INV_MMR_L2 Group divided by INV_MMR_L1 Group) for antibodies to rubella virus at Day 42; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANOVA; [statistical method as in outcome 2, analysis 1]; Adjusted GMC ratio = 0.93, 95% CI 2-sided [0.87 to 0.99]
Statistical Analysis 4: Comparison: INV_MMR_L2 Group vs INV_MMR_L3 Group; Adjusted GMC ratio (INV_MMR_L2 Group divided by INV_MMR_L3 Group) for antibodies to rubella virus at Day 42; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANOVA; [statistical method as in outcome 2, analysis 1]; Adjusted GMC ratio = 0.93, 95% CI 2-sided [0.87 to 0.99]
Statistical Analysis 5: Comparison: INV_MMR_L1 Group vs INV_MMR_L3 Group; Adjusted GMC ratio (INV_MMR_L3 Group divided by INV_MMR_L1 Group) for antibodies to rubella virus at Day 42; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANOVA; [statistical method as in outcome 2, analysis 1]; Adjusted GMC ratio = 1.00, 95% CI 2-sided [0.93 to 1.07]
Statistical Analysis 6: Comparison: INV_MMR_L2 Group vs INV_MMR_L3 Group; Adjusted GMC ratio (INV_MMR_L3 Group divided by INV_MMR_L2 Group) for antibodies to rubella virus at Day 42; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANOVA; [statistical method as in outcome 2, analysis 1]; Adjusted GMC ratio = 1.08, 95% CI 2-sided [1.01 to 1.15]

7. Primary Outcome: Percentage of Subjects With Anti-measles Virus Antibody Concentration Equal to or Above the Cut-off-value in Pooled MMR Groups
Description: Seroresponse was defined as post-vaccination anti-measles virus antibody concentration ≥200 mIU/mL among subjects who were seronegative (antibody concentration <150 mIU/mL) before vaccination. Criteria to demonstrate an acceptable immune response for INV_MMR in terms of seroresponse rates to measles virus at Day 42: The LL of 2-sided 95% CI for the seroresponse rate for the pooled INV_MMR lots is ≥90% for antibodies to measles virus.
Time Frame: At Day 42
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- INV_MMR Group: This group included subjects from INV_MMR _L1, INV_MMR _L2 and INV_MMR _L3 groups for whom pooled analysis was conducted in addition to lot-to-lot consistency.
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 3248 | 1137
Percentage of subjects
  Anti-measles ≥ 150 mIU/mL | 98.4 [97.9 to 98.8] | 98.1 [97.1 to 98.8]
  Anti-measles ≥ 200 mIU/mL | 98.2 [97.6 to 98.6] | 98.0 [97.0 to 98.7]
Statistical Analysis 1: Comparison: INV_MMR Group vs COM_MMR Group; Difference in percentage (INV_MMR Group minus COM_MMR Group) of subjects with anti-measles antibody concentration at Day 42; Test type: Non-Inferiority — The Lower Limit (LL) of 2-sided 95 % CI for the difference in seroresponse (INV_MMR Group minus COM_MMR Group) should be ≥-5% for antibodies to measles virus; Difference in seroresponse rate = 0.18, 95% CI 2-sided [-0.68 to 1.25] — Asymptotic standardized 95% CIs for the difference in seroresponse rate

8. Primary Outcome: Anti-measles Virus Antibody Concentrations in Pooled MMR Groups
Description: Antibody concentrations were expressed as GMCs in mIU/mL.
Time Frame: At Day 42
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 3248 | 1137
mIU/mL | 3017.4 [2923.9 to 3113.8] | 3074.4 [2911.0 to 3246.9]
Statistical Analysis 1: Comparison: INV_MMR Group vs COM_MMR Group; Adjusted GMC ratio (INV_MMR Group divided by COM_MMR Group) for antibodies to measles virus at Day 42; Test type: Non-Inferiority — The LL of the 2-sided 95% CI on GMC ratio (INV_MMR Group over COM_MMR Group) should be ≥0.67 for antibodies to measles virus; ANOVA; 95% CI for GMC ratio (INV_MMR over COM_ MMR) was computed using ANOVA (vaccine groups & country as fixed effects) on log-transformed concentrations; Adjusted GMC ratio = 0.98, 95% CI 2-sided [0.93 to 1.05]

9. Primary Outcome: Percentage of Subjects With Anti-mumps Virus Antibody Concentration Equal to or Above the Cut-off-value in Pooled MMR Groups
Description: Seroresponse was defined as post-vaccination anti-mumps virus antibody concentration ≥10 EU/mL among subjects who were seronegative (antibody concentrations <5 EU/mL) before vaccination.
Time Frame: At Day 42
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 3187 | 1107
Percentage of subjects
  Anti-mumps ≥ 5 EU/mL | 99.4 [99.1 to 99.6] | 99.3 [98.6 to 99.7]
  Anti-mumps ≥ 10 EU/mL | 98.4 [97.9 to 98.8] | 97.6 [96.5 to 98.4]
Statistical Analysis 1: Comparison: INV_MMR Group vs COM_MMR Group; Difference in percentage (INV_MMR Group minus COM_MMR Group) of subjects with anti-mumps antibody concentration at Day 42; Test type: Non-Inferiority — The LL of 2-sided 95 % CI for the difference in seroresponse (INV_MMR Group minus COM_MMR Group) should be ≥-5% for antibodies to mumps virus; Difference in seroresponse rate = 0.81, 95% CI 2-sided [-0.1 to 1.96] — Asymptotic standardized 95% CIs for the difference in seroresponse rate

10. Primary Outcome: Anti-mumps Virus Antibody Concentration in Pooled MMR Groups
Description: Antibody concentrations were expressed as GMCs in EU/mL.
Time Frame: At Day 42
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 3187 | 1107
EU/mL | 72.4 [70.4 to 74.5] | 69.1 [65.7 to 72.7]
Statistical Analysis 1: Comparison: INV_MMR Group vs COM_MMR Group; Adjusted GMC ratio (INV_MMR Group divided by COM_MMR Group) for antibodies to mumps virus at Day 42; Test type: Non-Inferiority — The LL of the 2-sided 95% CI on GMC ratio (INV_MMR Group over COM_MMR Group) should be ≥0.67 for antibodies to mumps virus; ANOVA; [statistical method as in outcome 8, analysis 1]; Adjusted GMC ratio = 1.05, 95% CI 2-sided [0.99 to 1.11]

11. Primary Outcome: Percentage of Subjects With Anti-rubella Virus Antibody Concentration Equal to or Above the Cut-off-value in Pooled MMR Groups
Description: Seroresponse was defined as post-vaccination anti-rubella virus antibody concentration ≥10 IU/mL among subjects who were seronegative (antibody concentrations <4 IU/mL) before vaccination. Criteria to demonstrate an acceptable immune response for INV_MMR in terms of seroresponse rates to rubella virus at Day 42: The LL of 2-sided 95% CI for the seroresponse rate for the pooled INV_MMR lots is ≥90% for antibodies to rubella virus.
Time Frame: At Day 42
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 3245 | 1135
Percentage of subjects
  Anti-rubella ≥ 4 IU/mL | 99.5 [99.2 to 99.7] | 99.6 [99.0 to 99.9]
  Anti-rubella ≥ 10 IU/mL | 97.3 [96.7 to 97.9] | 98.5 [97.6 to 99.1]
Statistical Analysis 1: Comparison: INV_MMR Group vs COM_MMR Group; Difference in percentage (INV_MMR Group minus COM_MMR Group) of subjects with anti-rubella antibody concentration at Day 42; Test type: Non-Inferiority — The LL of 2-sided 95 % CI for the difference in seroresponse (INV_MMR Group minus COM_MMR Group) should be ≥-5% for antibodies to rubella virus; Difference in seroresponse rate = -1.15, 95% CI 2-sided [-2.00 to -0.15] — Asymptotic standardized 95% CIs for the difference in seroresponse rate

12. Primary Outcome: Anti-rubella Virus Antibody Concentration in Pooled MMR Groups
Description: Antibody concentrations were expressed as GMCs in IU/mL.
Time Frame: At Day 42
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 3245 | 1135
IU/mL | 55.7 [54.2 to 57.3] | 64.0 [61.1 to 67.0]
Statistical Analysis 1: Comparison: INV_MMR Group vs COM_MMR Group; Adjusted GMC ratio (INV_MMR Group divided by COM_MMR Group) for antibodies to rubella virus at Day 42; Test type: Non-Inferiority — [test comment as in outcome 8, analysis 1]; ANOVA; [statistical method as in outcome 8, analysis 1]; Adjusted GMC ratio = 0.87, 95% CI 2-sided [0.83 to 0.92]

13. Secondary Outcome: Percentage of Subjects With an Anti-Varicella Zoster Virus (VZV) Antibody Concentration Equal to or Above the Cut-off Value in US Sub-cohort of Pooled MMR Groups
Description: Seroresponse was defined as post-vaccination anti-VZV antibody concentration ≥75 mIU/mL among subjects who were seronegative (antibody concentration <25 mIU/mL) before vaccination.
Time Frame: At Day 42
Population: ATP cohort for immunogenicity included subjects from US sub-cohort who received at least 1 MMR vaccine, were below the assay cut-off at pre-vaccination & with pre & post dose serology results available for at least 1 antigen of MMR, did not meet any elimination criteria up to Visit 2 blood sample & complied with post dose blood sample schedule
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 1492 | 540
Percentage of subjects
  Anti-VZV ≥ 25 mIU/mL | 99.7 [99.3 to 99.9] | 99.6 [98.7 to 100]
  Anti-VZV ≥ 75 mIU/mL | 92.2 [90.7 to 93.5] | 90.9 [88.2 to 93.2]
Statistical Analysis 1: Comparison: INV_MMR Group vs COM_MMR Group; In US sub-cohort: Difference in percentage (INV_MMR Group minus COM_MMR Group) of subjects with anti-VZV antibody concentration at Day 42; Test type: Non-Inferiority — The LL of 2-sided 95 % CI for the difference in seroresponse (pooled INV_MMR Group minus pooled COM_MMR Group) should be ≥-10% for antibodies to VZV; Difference in seroresponse rate = 1.30, 95% CI 2-sided [-1.31 to 4.29] — Asymptotic standardized 95% CIs for the difference in seroresponse rate

14. Secondary Outcome: Anti-VZV Virus Antibody Concentration in US Sub-cohort of Pooled MMR Groups
Description: Antibody concentrations were expressed as GMCs in mIU/mL.
Time Frame: At Day 42
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 1492 | 540
mIU/mL | 169.6 [164.3 to 175] | 167.2 [158.2 to 176.7]
Statistical Analysis 1: Comparison: INV_MMR Group vs COM_MMR Group; In US sub-cohort: Adjusted GMC ratio (INV_MMR Group divided by COM_MMR Group) for antibodies to VZV virus at Day 42; Test type: Non-Inferiority — The LL of the 2-sided 95% CI on GMC ratio (INV_MMR Group over COM_MMR Group) should be ≥0.67 for antibodies to VZV; ANOVA; [statistical method as in outcome 8, analysis 1]; Adjusted GMC ratio = 1.01, 95% CI 2-sided [0.95 to 1.08]

15. Secondary Outcome: Percentage of Subjects With an Anti-HAV Antibody Concentration Equal to or Above the Cut-off Value in US Sub-cohort of Pooled MMR Groups
Description: Percentage of subjects with an Anti-HAV antibody concentration equal to or above 15 mIU/mL were reported.
Time Frame: At Day 42
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 783 | 285
Percentage of subjects | 88.9 [86.5 to 91.0] | 87.4 [82.9 to 91.0]

16. Secondary Outcome: Anti-HAV Antibody Concentrations in US Sub-cohort of Pooled MMR Groups
Description: Antibody concentrations were expressed as GMCs in mIU/mL.
Time Frame: At Day 42
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 783 | 285
mIU/mL | 42.0 [39.3 to 44.8] | 42.4 [38.1 to 47.2]
Statistical Analysis 1: Comparison: INV_MMR Group vs COM_MMR Group; In US sub-cohort: Adjusted GMC ratio (INV_MMR Group divided by COM_MMR Group) for antibodies to HAV virus at Day 42; Test type: Non-Inferiority — The LL of the 2-sided 95% CI on GMC ratio (INV_MMR Group over COM_MMR Group) was ≥0.5 for antibodies to HAV virus; ANOVA; [statistical method as in outcome 8, analysis 1]; Adjusted GMC ratio = 0.98, 95% CI 2-sided [0.86 to 1.11]

17. Secondary Outcome: Anti-S.Pneumoniae Antibody Concentration in US Sub-cohort of Pooled MMR Groups
Description: Antibody concentrations were expressed as GMCs in microgram/Milliliter (µg/mL).
Time Frame: At Day 42
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 759 | 266
µg/mL
  anti-PnPS 1 antibody | 2.257 [2.121 to 2.402] | 2.425 [2.195 to 2.679]
  anti-PnPS 3 antibody: number analyzed (Participants) | 758 | 265
  anti-PnPS 3 antibody | 0.506 [0.481 to 0.533] | 0.496 [0.454 to 0.542]
  anti-PnPS 4 antibody: number analyzed (Participants) | 753 | 266
  anti-PnPS 4 antibody | 1.618 [1.518 to 1.725] | 1.872 [1.676 to 2.091]
  anti-PnPS 5 antibody: number analyzed (Participants) | 757 | 266
  anti-PnPS 5 antibody | 2.106 [1.991 to 2.228] | 2.280 [2.085 to 2.493]
  anti-PnPS 6A antibody | 5.840 [5.508 to 6.192] | 5.743 [5.233 to 6.304]
  anti-PnPS 6B antibody: number analyzed (Participants) | 758 | 266
  anti-PnPS 6B antibody | 5.872 [5.504 to 6.265] | 5.838 [5.239 to 6.505]
  anti-PnPS 7F antibody: number analyzed (Participants) | 758 | 266
  anti-PnPS 7F antibody | 3.691 [3.489 to 3.905] | 3.814 [3.484 to 4.176]
  anti-PnPS 9V antibody | 2.318 [2.183 to 2.461] | 2.282 [2.065 to 2.521]
  anti-PnPS 14 antibody: number analyzed (Participants) | 757 | 266
  anti-PnPS 14 antibody | 6.578 [6.155 to 7.029] | 7.053 [6.368 to 7.811]
  anti-PnPS 18C antibody: number analyzed (Participants) | 759 | 265
  anti-PnPS 18C antibody | 2.102 [1.973 to 2.241] | 2.217 [1.990 to 2.470]
  anti-PnPS 19A antibody: number analyzed (Participants) | 759 | 265
  anti-PnPS 19A antibody | 4.731 [4.461 to 5.017] | 4.821 [4.372 to 5.317]
  anti-PnPS 19F antibody | 4.251 [4.013 to 4.504] | 4.260 [3.872 to 4.687]
  anti-PnPS 23F antibody: number analyzed (Participants) | 742 | 256
  anti-PnPS 23F antibody | 2.198 [2.051 to 2.355] | 2.291 [2.025 to 2.592]
Statistical Analysis 1: Comparison: INV_MMR Group vs COM_MMR Group; In US sub-cohort: Adjusted GMC ratio (INV_MMR Group divided by COM_MMR Group) for anti-PnPS 1 antibody at Day 42; Test type: Non-Inferiority — The LL of the 2-sided 95% CI for GMC ratio (INV_MMR Group over COM_MMR Group) should be ≥0.5 for antibodies to for antibodies to PS serotypes; ANCOVA; 95% CI for GMC ratio (INV_MMR Group over the COM_MMR Group) was computed using an ANCOVA model: Adjustment for baseline concentration-pooled variance; Adjusted GMC ratio = 0.94, 95% CI 2-sided [0.85 to 1.05]
Statistical Analysis 2: Comparison: INV_MMR Group vs COM_MMR Group; In US sub-cohort: Adjusted GMC ratio (INV_MMR Group divided by COM_MMR Group) for anti-PnPS 3 antibody at Day 42; Test type: Non-Inferiority — [test comment as in outcome 17, analysis 1]; ANCOVA; [statistical method as in outcome 17, analysis 1]; Adjusted GMC ratio = 0.99, 95% CI 2-sided [0.91 to 1.08]
Statistical Analysis 3: Comparison: INV_MMR Group vs COM_MMR Group; In US sub-cohort: Adjusted GMC ratio (INV_MMR Group divided by COM_MMR Group) for anti-PnPS 4 antibody at Day 42; Test type: Non-Inferiority — [test comment as in outcome 17, analysis 1]; ANCOVA; [statistical method as in outcome 17, analysis 1]; Adjusted GMC ratio = 0.88, 95% CI [0.79 to 0.98]
Statistical Analysis 4: Comparison: INV_MMR Group vs COM_MMR Group; In US sub-cohort: Adjusted GMC ratio (INV_MMR Group divided by COM_MMR Group) for anti-PnPS 5 antibody at Day 42; Test type: Non-Inferiority — [test comment as in outcome 17, analysis 1]; ANCOVA; [statistical method as in outcome 17, analysis 1]; Adjusted GMC ratio = 0.92, 95% CI 2-sided [0.83 to 1.01]
Statistical Analysis 5: Comparison: INV_MMR Group vs COM_MMR Group; In US sub-cohort: Adjusted GMC ratio (INV_MMR Group divided by COM_MMR Group) for anti-PnPS 6A antibody at Day 42; Test type: Non-Inferiority — [test comment as in outcome 17, analysis 1]; ANCOVA; [statistical method as in outcome 17, analysis 1]; Adjusted GMC ratio = 1.01, 95% CI 2-sided [0.92 to 1.11]
Statistical Analysis 6: Comparison: INV_MMR Group vs COM_MMR Group; In US sub-cohort: Adjusted GMC ratio (INV_MMR Group divided by COM_MMR Group) for anti-PnPS 6B antibody at Day 42; Test type: Non-Inferiority — [test comment as in outcome 17, analysis 1]; ANCOVA; [statistical method as in outcome 17, analysis 1]; Adjusted GMC ratio = 0.98, 95% CI 2-sided [0.89 to 1.09]
Statistical Analysis 7: Comparison: INV_MMR Group vs COM_MMR Group; In US sub-cohort: Adjusted GMC ratio (INV_MMR Group divided by COM_MMR Group) for anti-PnPS 7F antibody at Day 42; Test type: Non-Inferiority — [test comment as in outcome 17, analysis 1]; ANCOVA; [statistical method as in outcome 17, analysis 1]; Adjusted GMC ratio = 0.94, 95% CI 2-sided [0.86 to 1.03]
Statistical Analysis 8: Comparison: INV_MMR Group vs COM_MMR Group; In US sub-cohort: Adjusted GMC ratio (INV_MMR Group divided by COM_MMR Group) for anti-PnPS 9V antibody at Day 42; Test type: Non-Inferiority — [test comment as in outcome 17, analysis 1]; ANCOVA; [statistical method as in outcome 17, analysis 1]; Adjusted GMC ratio = 0.99, 95% CI 2-sided [0.90 to 1.08]
Statistical Analysis 9: Comparison: INV_MMR Group vs COM_MMR Group; In US sub-cohort: Adjusted GMC ratio (INV_MMR Group divided by COM_MMR Group) for anti-PnPS 14 antibody at Day 42; Test type: Non-Inferiority — [test comment as in outcome 17, analysis 1]; ANCOVA; [statistical method as in outcome 17, analysis 1]; Adjusted GMC ratio = 0.91, 95% CI 2-sided [0.81 to 1.02]
Statistical Analysis 10: Comparison: INV_MMR Group vs COM_MMR Group; In US sub-cohort: Adjusted GMC ratio (INV_MMR Group divided by COM_MMR Group) for anti-PnPS 18C antibody at Day 42; Test type: Non-Inferiority — [test comment as in outcome 17, analysis 1]; ANCOVA; [statistical method as in outcome 17, analysis 1]; Adjusted GMC ratio = 0.92, 95% CI 2-sided [0.84 to 1.02]
Statistical Analysis 11: Comparison: INV_MMR Group vs COM_MMR Group; In US sub-cohort: Adjusted GMC ratio (INV_MMR Group divided by COM_MMR Group) for anti-PnPS 19A antibody at Day 42; Test type: Non-Inferiority — [test comment as in outcome 17, analysis 1]; ANCOVA; [statistical method as in outcome 17, analysis 1]; Adjusted GMC ratio = 0.97, 95% CI 2-sided [0.87 to 1.07]
Statistical Analysis 12: Comparison: INV_MMR Group vs COM_MMR Group; In US sub-cohort: Adjusted GMC ratio (INV_MMR Group divided by COM_MMR Group) for anti-PnPS 19F antibody at Day 42; Test type: Non-Inferiority — [test comment as in outcome 17, analysis 1]; ANCOVA; [statistical method as in outcome 17, analysis 1]; Adjusted GMC ratio = 0.96, 95% CI 2-sided [0.87 to 1.06]
Statistical Analysis 13: Comparison: INV_MMR Group vs COM_MMR Group; In US sub-cohort: Adjusted GMC ratio (INV_MMR Group divided by COM_MMR Group) for anti-PnPS 23F antibody at Day 42; Test type: Non-Inferiority — [test comment as in outcome 17, analysis 1]; ANCOVA; [statistical method as in outcome 17, analysis 1]; Adjusted GMC ratio = 0.95, 95% CI 2-sided [0.85 to 1.06]

18. Secondary Outcome: Number of Subjects With Any Solicited Local Adverse Events (AEs)
Description: Assessed solicited local AEs were pain, redness and swelling. Any = Occurrence of the symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 4-days (Days 0-3) post-vaccination period
Population: Total Vaccinated cohort (TVC) included all subjects with at least one vaccine administration of either INV_MMR or COM_MMR lots documented
Measure: Count of Participants; unit: Participants
Arm/Group | INV_MMR_L1 Group | INV_MMR_L2 Group | INV_MMR_L3 Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 1186 | 1175 | 1194 | 3555 | 1242
Participants
  Any Pain | 331 | 315 | 273 | 919 | 349
  Any Redness | 296 | 273 | 301 | 870 | 313
  Any Swelling | 116 | 99 | 103 | 318 | 133

19. Secondary Outcome: Number of Subjects With Any Solicited General AEs
Description: Assessed solicited general AEs were drowsiness, irritability and loss of appetite. Any = Occurrence of the symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 15-days (Days 0-14) post-vaccination period
Population: TVC included all subjects with at least one vaccine administration of either INV_MMR or COM_MMR lots documented
Measure: Count of Participants; unit: Participants
Arm/Group | INV_MMR_L1 Group | INV_MMR_L2 Group | INV_MMR_L3 Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 1190 | 1176 | 1200 | 3566 | 1243
Participants
  Any Drowsiness | 533 | 535 | 533 | 1601 | 586
  Any Irritability/fussiness | 764 | 729 | 765 | 2258 | 819
  Any Loss of appetite | 546 | 536 | 526 | 1608 | 548

20. Secondary Outcome: Number of Subjects Reporting Any Fever
Description: Any fever = Fever ≥ 38°C.
Time Frame: During the 43-days (Days 0-42) post-vaccination period
Population: TVC included all subjects with at least one vaccine administration of either INV_MMR or COM_MMR lots documented
Measure: Count of Participants; unit: Participants
Arm/Group | INV_MMR_L1 Group | INV_MMR_L2 Group | INV_MMR_L3 Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 1190 | 1176 | 1200 | 3566 | 1243
Participants | 404 | 422 | 418 | 1244 | 412

21. Secondary Outcome: Number of Subjects Reporting Any Rash
Description: Assessed were any localized or generalized rash, rash with fever, varicella-like rash, measles/rubella-like rash. Any = Occurrence of the symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 43-days (Days 0-42) post-vaccination period
Population: TVC included all subjects with at least one vaccine administration of either INV_MMR or COM_MMR lots documented
Measure: Count of Participants; unit: Participants
Arm/Group | INV_MMR_L1 Group | INV_MMR_L2 Group | INV_MMR_L3 Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 1190 | 1176 | 1200 | 3566 | 1243
Participants
  Any Localized or Generalized | 352 | 331 | 360 | 1043 | 378
  Any with fever | 106 | 123 | 118 | 347 | 104
  Any Varicella like | 87 | 78 | 85 | 250 | 85
  Any Measles/Rubella like | 71 | 88 | 76 | 235 | 77

22. Secondary Outcome: Number of Subjects Reporting Any MMR Specific Solicited AEs
Description: Assessed MMR specific solicited AEs were any suspected signs of meningism including febrile convulsions and parotid/salivary gland swelling. Any = Occurrence of the symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 43-days (Days 0-42) post-vaccination period
Population: TVC included all subjects with at least one vaccine administration of either INV_MMR or COM_MMR lots documented
Measure: Count of Participants; unit: Participants
Arm/Group | INV_MMR_L1 Group | INV_MMR_L2 Group | INV_MMR_L3 Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 1190 | 1176 | 1200 | 3566 | 1243
Participants
  Any febrile convulsion | 4 | 1 | 5 | 10 | 3
  Any parotid/salivary gland swelling | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Number of Subjects Reporting Any Unsolicited AEs
Description: Unsolicited adverse event (AE) was defined as any adverse event reported in addition to those solicited during the clinical study and also any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = Occurrence of the symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 43-days (Days 0-42) post-vaccination period
Population: TVC included all subjects with at least one vaccine administration of either INV_MMR or COM_MMR lots documented
Measure: Count of Participants; unit: Participants
Arm/Group | INV_MMR_L1 Group | INV_MMR_L2 Group | INV_MMR_L3 Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 1239 | 1232 | 1243 | 3714 | 1289
Participants | 615 | 633 | 609 | 1857 | 618

24. Secondary Outcome: Number of Subjects Reporting AEs of Specific Interest
Description: AEs of specific interest included new onset chronic disease (NOCD) (e.g., autoimmune disorders, asthma, type I diabetes, vasculitis, celiac disease, conditions associated with sub-acute or chronic thrombocytopenia and allergies) and AEs prompting emergency room (ER) visits.
Time Frame: From Day 0 through the end of study (Day 180)
Population: TVC included all subjects with at least one vaccine administration of either INV_MMR or COM_MMR lots documented
Measure: Count of Participants; unit: Participants
Arm/Group | INV_MMR_L1 Group | INV_MMR_L2 Group | INV_MMR_L3 Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 1239 | 1232 | 1243 | 3714 | 1289
Participants
  NOCDs | 40 | 39 | 49 | 128 | 48
  AEs prompting ER visits | 123 | 116 | 136 | 375 | 134

25. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity. Any SAE = Occurrence of SAE regardless of intensity grade or relation to vaccination.
Time Frame: From Day 0 through the end of study (Day 180)
Population: TVC included all subjects with at least one vaccine administration of either INV_MMR or COM_MMR lots documented
Measure: Count of Participants; unit: Participants
Arm/Group | INV_MMR_L1 Group | INV_MMR_L2 Group | INV_MMR_L3 Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 1239 | 1232 | 1243 | 3714 | 1289
Participants | 21 | 28 | 28 | 77 | 25

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: From Day 0 through the end of study (Day-180); Solicited local and general symptoms: During the 4-day (Day 0-3) and 15-days (Day 0-14) post-vaccination period; Unsolicited adverse events: During the 43-days (Day 0-42) post-vaccination period.
Description: The analysis of the solicited symptoms was based on the Total Vaccinated cohort which included only children/doses with documented safety data (i.e., symptom screen/sheet completed).
Arm/Group | INV_MMR_L1 Group | INV_MMR_L2 Group | INV_MMR_L3 Group | INV_MMR Group | COM_MMR Group
All-Cause Mortality (participants affected / at risk) | 0/1239 | 0/1232 | 0/1243 | 0/3714 | 0/1289
Serious Adverse Events (participants affected / at risk) | 21/1239 | 28/1232 | 28/1243 | 77/3714 | 25/1289
Other Adverse Events (participants affected / at risk) | 1089/1239 | 1053/1232 | 1090/1243 | 3232/3714 | 1138/1289
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INV_MMR_L1 Group (N=1239) | INV_MMR_L2 Group (N=1232) | INV_MMR_L3 Group (N=1243) | INV_MMR Group (N=3714) | COM_MMR Group (N=1289)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Milk allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 2 (2)
Bronchitis (Infections and infestations) | 3 (3) | 2 (2) | 3 (3) | 8 (8) | 2 (3)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Croup infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 2 (2)
Gastroenteritis adenovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Herpangina (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Mycoplasma infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neutropenic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 4 (4) | 2 (2)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 6 (6) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rotavirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (3) | 5 (5) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 4 (4) | 2 (2)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Finger amputation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INV_MMR_L1 Group (N=1239) | INV_MMR_L2 Group (N=1232) | INV_MMR_L3 Group (N=1243) | INV_MMR Group (N=3714) | COM_MMR Group (N=1289)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (6)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acquired phimosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Adenovirus infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 4 (4) | 6 (6) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 7 (7) | 7 (7) | 5 (5) | 19 (19) | 4 (4)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 4 (5)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Beta haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bilateral breast buds (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Bronchiolitis (Infections and infestations) | 2 (2) | 7 (7) | 7 (7) | 16 (16) | 6 (6)
Bronchitis (Infections and infestations) | 10 (10) | 12 (13) | 10 (11) | 32 (34) | 12 (13)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 3 (3) | 7 (7) | 2 (2)
Bullous impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 2 (3) | 1 (1) | 4 (5) | 2 (2)
Candida nappy rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 5 (5) | 0 (0)
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chemical poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cold agglutinins positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 26 (26) | 21 (21) | 39 (41) | 86 (88) | 32 (33)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 2 (2) | 9 (9) | 16 (16) | 8 (8)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 1 (1) | 5 (5) | 4 (4)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 33 (36) | 42 (42) | 38 (38) | 113 (116) | 36 (38)
Coxsackie viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Croup infectious (Infections and infestations) | 4 (4) | 11 (11) | 8 (8) | 23 (23) | 6 (6)
Crying (General disorders) | 4 (4) | 5 (7) | 2 (2) | 11 (13) | 4 (5)
Cyst (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 547 (548) | 537 (538) | 526 (528) | 1610 (1614) | 549 (550)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 4 (4) | 9 (9) | 3 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 5 (5) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 3 (4) | 4 (4) | 3 (4) | 10 (12) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 64 (71) | 58 (63) | 49 (55) | 171 (189) | 64 (68)
Diet noncompliance (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Drooling (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ear canal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 9 (9) | 14 (14) | 4 (4) | 27 (27) | 13 (13)
Ear injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 3 (3) | 3 (3) | 4 (4) | 10 (10) | 4 (4)
Ear swelling (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 5 (5)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Elbow deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterovirus infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 1 (1) | 7 (7) | 2 (2)
Epstein-barr virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Exaggerated startle response (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exanthema subitum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 5 (5) | 4 (4)
Eye inflammation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Febrile convulsion (Nervous system disorders) | 4 (4) | 1 (1) | 5 (5) | 10 (10) | 3 (3)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 5 (5) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 0 (0)
Food allergy (Immune system disorders) | 2 (2) | 2 (2) | 5 (6) | 9 (10) | 4 (4)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 27 (28) | 21 (21) | 35 (38) | 83 (87) | 31 (32)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 6 (6) | 6 (6) | 15 (15) | 6 (6)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 4 (4) | 3 (3)
Genital labial adhesions (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gingival hypertrophy (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gingival injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Gross motor delay (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 2 (2) | 3 (3) | 9 (9) | 14 (14) | 5 (5)
Head injury (Injury, poisoning and procedural complications) | 5 (5) | 6 (6) | 6 (6) | 17 (17) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1) | 5 (5) | 1 (1)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpangina (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypermetropia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 2 (2)
Immunisation reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 4 (4) | 1 (1) | 1 (1) | 6 (6) | 2 (2)
Infected bite (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 5 (5) | 1 (1) | 8 (8) | 10 (12)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 4 (4) | 5 (5) | 1 (1) | 10 (10) | 2 (2)
Injection site erosion (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Injection site erythema (General disorders) | 321 (331) | 294 (303) | 328 (334) | 943 (968) | 335 (341)
Injection site haematoma (General disorders) | 5 (6) | 1 (1) | 3 (3) | 9 (10) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Injection site induration (General disorders) | 3 (3) | 3 (3) | 2 (2) | 8 (8) | 3 (3)
Injection site mass (General disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Injection site nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 335 (336) | 316 (317) | 275 (277) | 926 (930) | 352 (352)
Injection site papule (General disorders) | 2 (2) | 2 (2) | 1 (1) | 5 (5) | 5 (5)
Injection site swelling (General disorders) | 127 (128) | 106 (107) | 113 (115) | 346 (350) | 139 (142)
Injection site vesicles (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 765 (775) | 730 (741) | 768 (775) | 2263 (2291) | 822 (838)
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 5 (5) | 0 (0) | 2 (2) | 7 (7) | 2 (2)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 7 (9) | 2 (2) | 10 (12) | 6 (6)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lice infestation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lid sulcus deepened (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0) | 4 (4) | 2 (2)
Lip injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 5 (5) | 5 (5) | 2 (2) | 12 (12) | 4 (4)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Middle insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Milk allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Nail avulsion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 11 (12) | 5 (5) | 26 (27) | 11 (11)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 74 (83) | 75 (82) | 74 (82) | 223 (247) | 65 (68)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 5 (5) | 0 (0)
Oral contusion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral mucosal eruption (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Otic examination normal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 80 (86) | 75 (79) | 62 (67) | 217 (232) | 86 (89)
Otitis media acute (Infections and infestations) | 8 (10) | 7 (7) | 13 (14) | 28 (31) | 9 (9)
Otitis media chronic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 20 (20) | 30 (30) | 14 (14) | 64 (64) | 23 (24)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 5 (5) | 7 (7) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Poor quality sleep (Nervous system disorders) | 4 (5) | 0 (0) | 1 (1) | 5 (6) | 1 (1)
Post-traumatic headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post-tussive vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prurigo (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 405 (406) | 422 (423) | 419 (419) | 1246 (1248) | 412 (412)
Radial head dislocation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ranula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 352 (352) | 331 (331) | 360 (360) | 1043 (1043) | 378 (378)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 4 (4) | 6 (6) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 8 (8) | 11 (12) | 9 (11) | 28 (31) | 7 (9)
Respiratory tract infection viral (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 4 (4) | 4 (4)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 46 (50) | 49 (55) | 38 (42) | 133 (147) | 41 (44)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 3 (3) | 8 (8) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 22 (23) | 23 (26) | 20 (21) | 65 (70) | 21 (22)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Roseola (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 0 (0)
Salivary gland enlargement (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Salivary gland pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Salmonellosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Scarlet fever (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (2) | 2 (2) | 0 (0) | 4 (4) | 1 (1)
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Secretion discharge (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (3) | 0 (0)
Sinusitis (Infections and infestations) | 9 (10) | 3 (3) | 4 (4) | 16 (17) | 3 (3)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin candida (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin warm (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Sleep disorder (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Sleep terror (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 534 (534) | 535 (535) | 533 (533) | 1602 (1602) | 586 (586)
Speech disorder developmental (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1) | 5 (5) | 1 (1)
Strabismus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Streptococcal infection (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 5 (5) | 3 (3)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Superficial injury of eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tearfulness (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Teething (Gastrointestinal disorders) | 91 (114) | 92 (106) | 77 (92) | 260 (312) | 95 (114)
Terminal insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 21 (22) | 9 (10) | 9 (11) | 39 (43) | 15 (16)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 4 (6) | 0 (0) | 1 (1) | 5 (7) | 6 (7)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 106 (117) | 124 (132) | 122 (132) | 352 (381) | 122 (129)
Urinary tract disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 1 (1) | 1 (1) | 3 (4) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1) | 1 (1) | 4 (6) | 0 (0)
Vaginal mucosal blistering (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Viral diarrhoea (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Viral infection (Infections and infestations) | 15 (15) | 21 (22) | 23 (26) | 59 (63) | 15 (15)
Viral pharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 4 (4) | 1 (1)
Viral rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Viral tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3) | 4 (4) | 10 (10) | 3 (3)
Vomiting (Gastrointestinal disorders) | 38 (39) | 35 (38) | 34 (38) | 107 (115) | 43 (46)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 6 (6) | 6 (6) | 14 (15) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.